CLINICAL TRIAL: NCT03819725
Title: Monitoring of Postprandial Glycemic Variability in Healthy Young Infants
Acronym: IGVM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Principal Investigator, Michael Hauschild, Dr. Michael Hauschild, MD, University of Lausanne Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CER-VD / 2017-02090
Record Dates: First submitted 2018-12-23; First posted 2019-01-28 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Infant Conditions; Glucose Intolerance
Keywords: Glucose variation; Infant; Nutrition; interstitial glucose variation
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glucose monitoring (Other): FreeStyle® Libre Pro Interstitial Glucose Meter will be applied after skin preparation with anesthetic cream (Emla® ) and glucose measurements will be monitored during 2-5 days. Oral food intake will be recorded.
  Interventions: Device: Glucose monitoring

INTERVENTIONS:
Device: Glucose monitoring — FreeStyle® Libre Pro Interstitial Glucose Meter will be applied after skin preparation with anesthetic cream (Emla®) . Interstitial glucose measurements will be recorded during 2-5 days and during meals.

SUMMARY:
To measure and quantify the postprandial glucose variations in response to a meal in the healthy 6-12 months old child and correlate this response with the composition of this meal.

DETAILED DESCRIPTION:
14 full-term infants (boys and girls) aged six to twelve months and fed a diversified diet including infant formula, solid foods such as mixed meat and vegetable preparation or marketed preparations will be recruited. Children will be recruited in the Lausanne Childrens hospital and only be included in the study whenin good general health.

FreeStyle® Libre Pro Interstitial Glucose Meter will be applied on the last day before discharge from the hospital after skin preparation with anesthetic cream (Emla®) during hospitalization and measurements will be recorded during 2-5 days.

It is not intended to measure capillary or venous blood glucose levels during this study. However, if blood is collected during hospitalization, blood glucose will be measured in parallel with the interstitial glucose measured with the device.

The child will follow his usual diet without modifications. The amount of food consumed by the child as well as the length of the meals will be recorded by the parents. For meals made by the parents they will be asked to keep a sample not seen to analyze their carbohydrate content. The total carbohydrate content will be measured .

ELIGIBILITY:
Inclusion Criteria:

* Term infants (boys and girls)
* 6 to 12 months old
* In good general health
* Nourished with diverse nutrition including infant formula, solid foods such as mixed meat and vegetable preparation or marketed preparations
* Infant child: if the child is breastfed partially, it can be included in the study. In this case, only samples of a food supplement will be collected for evaluation of the composition.
* Hospitalized at the Lausanne Children's Hospital for non-severe reasons that do not affect or suspect to affect glucose metabolism
* Measures of feeding (time and compositions with samples) feasible for 3 consecutive days by the parents at home

Exclusion Criteria:

* Child born premature
* One or both parents with type 2 diabetes or gestational diabetes
* Child totally breastfed
* Chronic skin condition such as eczema, excessive dryness.
* Allergy known to adhesive plaster
* Infectious diseases affecting the skin (eg chickenpox, scarlet fever,)
* disorders of cutaneous microcirculation
* Infants suffering from diseases affecting nutrition or digestion (diarrheal gastroenteritis) and children undergoing antibiotic treatment that may affect gastrointestinal absorption
* Magnetic Resonance Imaging (MRI), Computed Tomography (CT), or Diathermy Therapy

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Prandial glucose variations | up to 5 days
  Change of preprandial to postprandial glucose measurements, expressed in mmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hauschild, MF, Principal Investigator — CHUV
Locations (1):
- Pediatric Endocrinology, Diabetology and Obesity Unit, Service of Pediatrics, Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided